CLINICAL TRIAL: NCT00306917
Title: A Prospective, Randomized Study of Summit™ Porocoat® Versus Summit™ DuoFix™ HA in Cementless Total Hip Arthroplasty
Brief Title: Clinical Study Comparing Two Implant Surface Finishes in Patients Undergoing Cementless Total Hip Replacement
Acronym: SPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to limited enrollment and follow up.
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Avascular Necrosis; Acute Fracture
Keywords: Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DuoFix HA
  Interventions: Device: non-coated femoral hip stem
- 2 (Active Comparator): Porocoat porous coated
  Interventions: Device: coated femoral hip stem

INTERVENTIONS:
Device: non-coated femoral hip stem — total hip replacement
  Other Names: Summit DuoFix HA hip stem
  Arms: 1
Device: coated femoral hip stem — total hip replacement
  Other Names: Summit Porocoated porous coated hip stem.
  Arms: 2

SUMMARY:
Prospective, randomized study of Summit Porocoat versus Summit DuoFix HA in total hip arthroplasty

DETAILED DESCRIPTION:
Hydroxyapatite (HA) is a bioactive ceramic that resembles the natural inorganic mineral content of bone, and as such is a highly osteoconductive material. The purpose of this study is to compare an HA coated and uncoated prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip replacement
* Patient age less than or equal to 75
* Sufficient bone stock to support prosthesis

Exclusion Criteria:

* Previous hip replacement
* Significant angular/bony deformity
* Active joint sepsis
* Metal allergy
* Renal transplant
* Psychosocial disease
* Neurological disease/musculoskeletal disease that may affect weight-bearing

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2002-11-01 (Actual); Primary Completion 2009-01-29 (Actual); Study Completion 2009-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Fisher, MD, Principal Investigator — Orthopaedics Indianapolis; J W Mesko, MD, Principal Investigator — Michigan Orthopaedics Center; Paul Perona, MD, Principal Investigator — St Margaret's Hospital Family Orthopaedics; Stephan B Lowe, MD, Principal Investigator — Orthopaedic Specialists of the Carolinas; Donald L Pomeroy, MD, Principal Investigator — Pomeroy & Reddy; Nithin Reddy, MD, Principal Investigator — Pomeroy & Reddy
Locations (1):
- DePuy Orthopaedics, Warsaw, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in September 2002 and ended June 2006. Study subjects were recruited and enrolled in medical clinics by orthopaedic surgeons at eight investigational sites. Each site could enroll a maximum of 50 subjects. Recruitment was based on the inclusion and exclusion criteria as indicated in the study protocol.
Pre-assignment Details: Immediately before surgery, the implant type was determined according to the randomization schedule. Enrolled subjects may have been excluded from the trial before assignment to the study arm based upon results of pre-operative clinical evaluations and radiographs that would exclude a subject based on exclusion criteria in the study protocol.
Groups:
- DuoFix HA: The Summit™ DuoFix™ HA stems are primary, cementless hip implants. Summit™ cementless stems feature 3°-tapered body geometry to enhance fit, and are manufactured from forged titanium alloy. The Summit™ cementless stems are designed to load the femur toward the upper part of the stem, and therefore the Porocoat® porous coating is applied only to the upper body of the stem. The DuoFix™ HA stem also has a thin coating of hydroxyapatite on this porous-coated surface. This HA coating is only 35 microns thick, so the optimum pore size is maintained. The lower portion of the stem has a grit-blasted surface, which promotes bone on-growth and the polished bullet-tip prevents end-stem loading.
- Porocoat Porous Coated: The Summit™ Porocoat® stems are primary, cementless hip implants that a feature 3°-tapered body geometry to enhance fit, and are manufactured from forged titanium alloy. The Summit™ cementless stems are designed to load the femur toward the upper part of the stem, and therefore the Porocoat® porous coating is applied only to the upper body of the stem. The lower portion of the stems has a grit-blasted surface, which promotes bone on-growth and the polished bullet-tip prevents end-stem loading.
Period: Overall Study
Arm/Group | DuoFix HA | Porocoat Porous Coated
Started | 121 (400 subjects were to be followed for 5 years; due to slow enrollment study closed early with 245.) | 124 (400 subjects were to be followed for 5 years; due to slow enrollment study closed early with 245.)
Postoperative to 6 Month Follow up | 93 | 100
12 Month Follow | 86 | 94
24 Month Follow up | 60 | 71
36 Month Follow up | 56 | 42
48 Month Follow up | 29 | 22
60 Month Follow up | 13 | 15
Completed | 13 | 15
Not Completed | 108 | 109

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DuoFix HA | Porocoat Porous Coated | Total
Number analyzed (Participants) | 121 | 124 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.2) | 63.2 (9.2) | 63.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 64 | 131
  Male | 54 | 60 | 114
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 121 | 124 | 245

OUTCOME MEASURES:

1. Secondary Outcome: Medical Imaging as a Secondary Outcome Inclusive of All Post-operative Intervals for All Participants at Study Closure.
Description: Medical imaging as a secondary outcome inclusive of all post-operative intervals for all participants at study closure. This measure is a percentage of the overall Participants with a specific radiographic outcome. Measurements were made by an Independent Radiographic Reviewer (IRR) and include assessments made based on protocol defined radiographic success criteria that includes Subsidence (10 mm), Osseointegration, Radiolucency > 2 mm in any zone, Complete Circumferential Radiolucencies, Spot-Welds (AP View) p < .10, Spot-Welds (Lateral View) p < .10, Cortical Hypertrophy (AP View), Cortical Hypertrophy (Lateral View)
Time Frame: Postoperative, 6, 12, 24, 36, 48 and 60 months
Measure: Number; unit: Percentage of Participants Analyzed
Arm/Group | DuoFix HA | Porocoat Porous Coated
Number analyzed (Participants) | 121 | 124
Percentage of Participants Analyzed
  Subsidence (10 mm) | 1 | 0
  Osseointegration | 82 | 80
  Radiolucency > 2 mm in any zone | 0 | 0
  Complete Circumferential Radiolucencies | 0 | 0
  Spot-Welds (AP View) p < .10 | 23 | 14
  Spot-Welds (Lateral View) p < .10 | 8 | 3
  Cortical Hypertrophy (AP View) | 12 | 12
  Cortical Hypertrophy (Lateral View) | 3 | 4

2. Primary Outcome: Harris Hip Score (HHS)
Description: The Harris Hip scoring system assigns a numeric value to responses from patients and assessments made by a surgeon. A score of 90-100 is excellent, 80-90 is good, 70-80 is fair, 60-69 is poor, and 60 or below is failed. The patient records the following: pain level, need for assistance when walking, presence of a limp, distance able to walk, ability to put on shoes and socks, climb stairs, use public transportation and the length of time one is able to comforatably sit in a chair are all scored. The doctor assesses patient hip function by testing flexion, extension, adduction and abduction.
Time Frame: Preoperative, 6, 12, 24, 36, 48, and 60 months
Population: Before the first interval there were five missing HHS scores for the DuoFix arm and four missing HHS scores for the Porocoat Porous Coated arm. At the final interval (60 months), there were eleven subjects in the DuoFix arm with complete HHS scores and there were fourteen subjects in the Porocoat Porous Coated arm with complete HHS scores.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DuoFix HA | Porocoat Porous Coated
Number analyzed (Participants) | 121 | 124
Units on a scale
  Preoperative HHS | 49.9 (13.4) | 51.2 (14.0)
  Postoperative to 6 Month HHS | 90.2 (10.3) | 91.6 (8.3)
  12 Month HHS | 92.8 (7.9) | 92.3 (11.6)
  24 Month HHS | 93.3 (7.8) | 93.5 (9.7)
  36 Month HHS | 94.0 (8.5) | 93.8 (9.4)
  48 Month HHS | 91.8 (12.2) | 95.5 (10.5)
  60 Month HHS | 93.8 (7.9) | 93.6 (7.8)

ADVERSE EVENTS:
Arm/Group | DuoFix HA | Porocoat Porous Coated
Serious Adverse Events (participants affected / at risk) | 3/121 | 4/124
Other Adverse Events (participants affected / at risk) | 6/121 | 7/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DuoFix HA (N=121) | Porocoat Porous Coated (N=124)
Cardiovascular Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dislocation (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection: Deep (Infections and infestations) | 1 (1) | 1 (1)
Infection: Superficial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Liner failure: dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DuoFix HA (N=121) | Porocoat Porous Coated (N=124)
Blood Loss Anemia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
The protocol called for 400 subjects to be followed for 5 years, but due to slow enrollment the study closed early. 245 subjects were enrolled & study endpoint was modified to 2 years. Enrollment closed on June 30, 2006; study closed on Jan 29, 2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less